CLINICAL TRIAL: NCT00566046
Title: Prospective, Randomized, Double-blind Study Assessing the Effects of Levetiracetam Compared to Placebo in the Prevention of Early Epileptic Seizures and Late Epilepsy in Patients With Severe Traumatic Brain Injury
Brief Title: Prevention of Post-traumatic Seizures With Levetiracetam
Acronym: TRACK
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision because of to small enrollment
Sponsor: Rennes University Hospital (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EudraCT: 2006-006518-13; CIC0203/60 (Other: Rennes University Hospital); LOC/06-06 (Other: Rennes University Hospital)
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Epilepsy, Post-Traumatic
MeSH Terms: conditions — Epilepsy, Post-Traumatic | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levetiracetam (Experimental)
  Interventions: Drug: Levetiracetam
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levetiracetam — 1500 mg/day orally until the first episode of late epilepsy for a maximum duration of 3 months
  Other Names: Keppra
  Arms: Levetiracetam
Drug: Placebo — 1500 mg/day orally until the first episode of late epilepsy for a maximum duration of 3 months
  Arms: Placebo

SUMMARY:
Post-traumatic seizures can appear frequently after a severe traumatic brain injury. Two types of seizures are usually identified: early seizures during the week following the trauma and late epilepsy afterward. Several antiepileptic drugs are usually used to prevent early seizures but no treatment has demonstrated any preventive effect against late epilepsy. Levetiracetam is an antiepileptic drug usually used for the treatment of epileptic patients and has pharmacologic properties that could also be interesting for the prevention of post-traumatic epilepsy.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years old
2. Patient with severe brain injury defined as follow:

   * Initial Glasgow Coma score (assessed on the scene of the accident) <= 8 related to the brain injury
   * Stage 2 to 4 on the TDM US TCDB classification
3. Initial brain CT scan performed within 48 hours after hospital admission
4. Either a male or a nonpregnant, non-lactating female who is using adequate contraceptive method (a urine laboratory pregnancy test must be negative at baseline)
5. Written informed consent from the patient's next-of-kin. If no relative is present as the time of inclusion, the patients will be included according to the emergency procedure

Exclusion Criteria:

1. Isolated extradural hematoma
2. Medical decision to limit patient's care (terminal stage of a cancer, hematological malignancies, HIV, etc.)
3. Current participation in an other protocol or within one month before study entry
4. Previous treatment with Levetiracetam
5. Patient's follow-up judged to be difficult by the investigator
6. Known allergy to either Levetiracetam or products derived from pyrrolidone or one of its excipients
7. Epileptic patient treated or not (except patients treated with benzodiazepines who can be included in this protocol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Time to early epileptic seizures (<= 8 days) and late epilepsy (from day 9 to 1 year) in patients with severe traumatic brain injury | one year

SECONDARY OUTCOMES:
Rate of early seizures and of late epilepsy; treatment effects according to the patient's severity, the TDM US Traumatic Coma Data Bank, and the number of regions traumatized; safety of Levetiracetam | One year
Global prognosis (Glasgow Outcome Scale) | 3 months, 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Biraben, MD, Principal Investigator — Rennes University Hospital; Bruno Laviolle, MD, Study Chair — Rennes University Hospital
Locations (15):
- France (15):
  - Neurologie - CHU Angers, Angers
  - Neurology - CHU Bordeaux, Bordeaux
  - Neurologie - CHU Caen, Caen
  - Neurochirurgie-CHU Grenoble, Grenoble
  - Neurology - CHU Rennes, Grenoble
  - Neurophysiologie Clinique - CHU Lille, Lille
  - Neurophysiologie clinique - CHU Lyon (Hôpital neurologique), Lyon
  - Beurophysiologie clinique - CHU Marseille, Marseille
  - Epileptologie - CHU Montpellier, Montpellier
  - Neurologie - CHU Nancy, Nancy
  - Neurochirurgie-Paris Saint Anne, Paris
  - Neurologie - CHU Rennes, Rennes
  - Explorations Fonctionnelles Neurologiques - CHU Nantes, Rennes
  - Neurologie - CHU Rouen, Rouen
  - Neurologie - CHU Tours Hopital Trousseau, Tours